CLINICAL TRIAL: NCT01011491
Title: Efficacy of Medifast's 5 & 1 Program Compared to a Food-based Diet After a Period of Weight Loss and Weight Maintenance
Brief Title: Comparison of Medifast's 5 & 1 Plan to a Food-based Plan of Equal Calories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medifast, Inc. (Industry)
Responsible Party: Lisa M. Davis, PhD, PA-C, CNS, LDN/ Vice President, Research & Development, Medifast, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED014; 20080292 (Other: Western Institutional Review Board)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; meal replacements; inflammation; oxidative stress; visceral fat
MeSH Terms: conditions — Obesity; Weight Loss; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medifast 5 & 1 Plan (Experimental): Medifast's 5 & 1 Plan is a meal replacement plan for weight loss and weight maintenance.
  Interventions: Other: Medifast 5 & 1 Plan for weight loss and weight maintenance
- Food-based (Active Comparator): The food-based arm followed a meal plan of self-selected foods that provided the same number of calories as the Medifast 5 & 1 plan.
  Interventions: Other: Food-based diet plan for weight loss and weight maintenance

INTERVENTIONS:
Other: Medifast 5 & 1 Plan for weight loss and weight maintenance — Medifast's 5 & 1 Plan is a meal replacement program for weight loss that uses 5 Medifast meals and 1 self-prepared meal. The weight maintenance plan incorporates 3-5 Medifast meals as well as a certain amount of food from all other food groups.
  Arms: Medifast 5 & 1 Plan
Other: Food-based diet plan for weight loss and weight maintenance — The food-based group was provided a meal plan for weight loss based on the guidelines of the USDA Food Guide Pyramid providing the same number of calories as the Medifast 5 & 1 Plan. Weight maintenance calories were calculated and participants were provided meal plans from the USDA Food Guide Pyramid.
  Arms: Food-based

SUMMARY:
Portion-controlled meal replacements have been shown to be an effective weight control strategy in overweight and obese individuals. Thus, the investigators plan to evaluate the effect of Medifast's 5 & 1 program compared to an food-based diet plan of equal calories on the following indices: weight loss and maintenance of weight loss, satiety during weight loss, changes in biochemical markers of inflammation and oxidative stress following weight loss, and compliance and retention rates.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females (age between 18 and 65)
* Obese (BMI >=30.0 kg/m2 and <50.0 kg/m2)
* Non-smokers
* No known food allergies to wheat, gluten, soy or nuts
* <14 alcoholic beverages per week
* Willing and able to give informed consent
* Not currently using appetite-affecting medications (e.g SSRIs, steroids, Ritalin)
* Not pregnant or lactating
* Primary care physician's permission for weight loss, normal labs and electrocardiogram (EKG) within past 1 year

Exclusion Criteria:

* Actively dieting
* Eating Attitudes Test (EAT) > 30
* Chronic uncontrolled health problems (not including obesity or diabetes)
* Pacemaker or other internal electronic medical device
* Schizophrenia, history of bipolar disorder, current Major Depressive Disorder
* Dependence on alcohol or sedative-hypnotic drugs (e.g. benzodiazepines)
* Cognitive impairment severe enough to preclude informed consent
* Taking weight loss or appetite-suppressant medications
* Taking appetite affecting medications (e.g. SSRIs, steroids, Ritalin)
* Food allergies to wheat, gluten, soy, or nuts
* Pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Weight change (in kilograms) from week 0 | 16 weeks

SECONDARY OUTCOMES:
Satiety using a visual analog scale | 16 weeks
Change in Inflammation represented by C-reactive protein | 16 and 40 weeks
Change in Oxidative Stress represented by urine lipid peroxides | 16 and 40 weeks
Blood Pressure change | 16 and 40 weeks
Change in Pulse | 16 and 40 weeks
Maintenance of weight lost during the 16 week weight loss phase expressed as weight regained from week 16 to week 40 (in kilograms) | 24 weeks
Change in percent body fat (a measure representing a change in body composition) | 16 and 40 weeks
Change in Blood lipids | 16 and 40 weeks
Change in lean muscle mass (a measure representing change in body composition) | 16 and 40 weeks
Change in Waist circumference (a measure representing change in body composition) | 16 and 40 weeks
Change in Visceral Fat Rating (a measure representing change in body composition) | 16 and 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Davis, PhD, PA-C, Principal Investigator — Medifast, Inc.
Locations (1):
- Medifast, Inc., Owings Mills, Maryland, United States

REFERENCES:
- [Background] Thearle M, Aronne LJ. Obesity and pharmacologic therapy. Endocrinol Metab Clin North Am. 2003 Dec;32(4):1005-24. doi: 10.1016/s0889-8529(03)00066-5. PMID 14711072
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] Gale SM, Castracane VD, Mantzoros CS. Energy homeostasis, obesity and eating disorders: recent advances in endocrinology. J Nutr. 2004 Feb;134(2):295-8. doi: 10.1093/jn/134.2.295. PMID 14747663
- [Background] de Ferranti S, Rifai N. C-reactive protein and cardiovascular disease: a review of risk prediction and interventions. Clin Chim Acta. 2002 Mar;317(1-2):1-15. doi: 10.1016/s0009-8981(01)00797-5. PMID 11814453
- [Background] Festi D, Colecchia A, Sacco T, Bondi M, Roda E, Marchesini G. Hepatic steatosis in obese patients: clinical aspects and prognostic significance. Obes Rev. 2004 Feb;5(1):27-42. doi: 10.1111/j.1467-789x.2004.00126.x. PMID 14969505
- [Background] Abbott RD, Ross GW, White LR, Nelson JS, Masaki KH, Tanner CM, Curb JD, Blanchette PL, Popper JS, Petrovitch H. Midlife adiposity and the future risk of Parkinson's disease. Neurology. 2002 Oct 8;59(7):1051-7. doi: 10.1212/wnl.59.7.1051. PMID 12370461
- [Background] Heymsfield SB, van Mierlo CA, van der Knaap HC, Heo M, Frier HI. Weight management using a meal replacement strategy: meta and pooling analysis from six studies. Int J Obes Relat Metab Disord. 2003 May;27(5):537-49. doi: 10.1038/sj.ijo.0802258. PMID 12704397
- [Background] Visser M, Bouter LM, McQuillan GM, Wener MH, Harris TB. Elevated C-reactive protein levels in overweight and obese adults. JAMA. 1999 Dec 8;282(22):2131-5. doi: 10.1001/jama.282.22.2131. PMID 10591334
- [Background] Yudkin JS, Stehouwer CD, Emeis JJ, Coppack SW. C-reactive protein in healthy subjects: associations with obesity, insulin resistance, and endothelial dysfunction: a potential role for cytokines originating from adipose tissue? Arterioscler Thromb Vasc Biol. 1999 Apr;19(4):972-8. doi: 10.1161/01.atv.19.4.972. PMID 10195925
- [Background] Tchernof A, Nolan A, Sites CK, Ades PA, Poehlman ET. Weight loss reduces C-reactive protein levels in obese postmenopausal women. Circulation. 2002 Feb 5;105(5):564-9. doi: 10.1161/hc0502.103331. PMID 11827920
- [Background] Furukawa S, Fujita T, Shimabukuro M, Iwaki M, Yamada Y, Nakajima Y, Nakayama O, Makishima M, Matsuda M, Shimomura I. Increased oxidative stress in obesity and its impact on metabolic syndrome. J Clin Invest. 2004 Dec;114(12):1752-61. doi: 10.1172/JCI21625. PMID 15599400
- [Background] Stefanovic A, Kotur-Stevuljevic J, Spasic S, Bogavac-Stanojevic N, Bujisic N. The influence of obesity on the oxidative stress status and the concentration of leptin in type 2 diabetes mellitus patients. Diabetes Res Clin Pract. 2008 Jan;79(1):156-63. doi: 10.1016/j.diabres.2007.07.019. Epub 2007 Sep 11. PMID 17850913
- [Background] Vincent HK, Morgan JW, Vincent KR. Obesity exacerbates oxidative stress levels after acute exercise. Med Sci Sports Exerc. 2004 May;36(5):772-9. doi: 10.1249/01.mss.0000126576.53038.e9. PMID 15126709
- [Background] Ashley JM, Herzog H, Clodfelter S, Bovee V, Schrage J, Pritsos C. Nutrient adequacy during weight loss interventions: a randomized study in women comparing the dietary intake in a meal replacement group with a traditional food group. Nutr J. 2007 Jun 25;6:12. doi: 10.1186/1475-2891-6-12. PMID 17592648
- [Background] Ditschuneit HH, Flechtner-Mors M. Value of structured meals for weight management: risk factors and long-term weight maintenance. Obes Res. 2001 Nov;9 Suppl 4:284S-289S. doi: 10.1038/oby.2001.132. PMID 11707555
- [Background] Egger GJ. Are meal replacements an effective clinical tool for weight loss?--a clarification. Med J Aust. 2006 Jun 5;184(11):591. doi: 10.5694/j.1326-5377.2006.tb00399.x. No abstract available. PMID 16768675
- [Background] Ball SD, Keller KR, Moyer-Mileur LJ, Ding YW, Donaldson D, Jackson WD. Prolongation of satiety after low versus moderately high glycemic index meals in obese adolescents. Pediatrics. 2003 Mar;111(3):488-94. doi: 10.1542/peds.111.3.488. PMID 12612226
- [Derived] Davis LM, Coleman C, Kiel J, Rampolla J, Hutchisen T, Ford L, Andersen WS, Hanlon-Mitola A. Efficacy of a meal replacement diet plan compared to a food-based diet plan after a period of weight loss and weight maintenance: a randomized controlled trial. Nutr J. 2010 Mar 11;9:11. doi: 10.1186/1475-2891-9-11. PMID 20222968